CLINICAL TRIAL: NCT03854708
Title: Effect of Pancreatic Polypeptide on Intragastric Pressure and Satiety During Nutrient Drink Infusion
Brief Title: Effect of Pancreatic Polypeptide on Gastric Motor Function and Food Intake in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PP and gastric motility
Record Dates: First submitted 2019-02-01; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-01

CONDITIONS: Hunger
Keywords: gastric accommodation; gastric emptying; hunger; satiety; nutrient tolerance
MeSH Terms: interventions — Pancreatic Polypeptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 pmol/kg*min pancreatic polypeptide (Experimental): 3 pmol/kg*min of pancreatic polypeptide was intravenously infused.
  Interventions: Drug: 3 pmol/kg*min pancreatic polypeptide
- 10 pmol/kg*min pancreatic polypeptide (Experimental): 10 pmol/kg*min of pancreatic polypeptide was intravenously infused.
  Interventions: Drug: 10 pmol/kg*min pancreatic polypeptide
- Placebo (Placebo Comparator): 0.9 % saline solution was intravenously infused.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3 pmol/kg*min pancreatic polypeptide — PP 3 pmol/kg*min was intravenously infused 30 minutes before the meal until the end of the meal. For this purpose, a cannula was inserted into the subjects' forearm vein. Human PP (CS Bio, Menlo Park, USA) was dissolved in a 0.9 % saline solution containing 5 % albumin to reduce absorption of PP to the syringe and tubing.
  Other Names: Pancreatic polypeptide
  Arms: 3 pmol/kg*min pancreatic polypeptide
Drug: 10 pmol/kg*min pancreatic polypeptide — PP 10 pmol/kg*min was intravenously infused 30 minutes before the meal until the end of the meal. For this purpose, a cannula was inserted into the subjects' forearm vein. Human PP (CS Bio, Menlo Park, USA) was dissolved in a 0.9 % saline solution containing 5 % albumin to reduce absorption of PP to the syringe and tubing.
  Other Names: Pancreatic polypeptide
  Arms: 10 pmol/kg*min pancreatic polypeptide
Drug: Placebo — Placebo (saline solution) was intravenously infused 30 minutes before the meal until the end of the meal. For this purpose, a cannula was inserted into the subjects' forearm vein. The placebo consists of a 0.9 % saline solution containing 5 % albumin.
  Arms: Placebo

SUMMARY:
The investigators want to observe whether different doses of pancreatic polypeptide infusions influence gastric accommodation (measured as intragastric pressure changes during a liquid meal infusion), gastric emptying and food intake.

DETAILED DESCRIPTION:
As pancreatic polypeptide (PP) influences food behavior in humans, our research group suggests a role via the the gastric accommodation or gastric emptying. Twelve healthy volunteers participated in this single blind, placebo-controlled, crossover trial. An infusion catheter and a manometry probe were positioned in the stomach. After a 15 min stabilization period, saline (placebo), PP 3 pmol/kg*min or PP 10 pmol/kg*min were intravenously infused. Thirty min after the condition, an intragastric nutrient drink (ND) infusion (60 ml/min) started until the volunteer felt maximal satiated. GE was evaluated using the 13C breath test during the 6 hours following the ND infusion. Satiation and hunger were scored on a visual analog scale every 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 65 years of age.
* Women of child-bearing potential agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject is under age of legal consent, pregnant or breastfeeding.
* Subject has current symptoms or a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies.
* Subject has a significant heart, lung, liver or kidney disease.
* Subject has any history of a neurological disorder. Subject has a history of abdominal surgery. Those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate.
* History or current use of drugs that can affect glycaemia, gastrointestinal function, motility or sensitivity or gastric acidity.
* History or current use of centrally acting medication, including antidepressants, antipsychotics and/or benzodiazepines (in the last year before screening visit).
* Subject consumes excessive amounts of alcohol, defined as >14 units per week for females and > 21 units per week for males.
* Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
* High caffeine intake (> 500 ml coffee daily or equivalent).
* Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.
* Recent participation (<30 days) or simultaneous participation in another clinical study.
* Subjects with lactose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2011-03-08 (Actual); Study Completion 2011-03-08 (Actual)

PRIMARY OUTCOMES:
The effect of different doses of pancreatic polypeptide infusion on the gastric accommodation (intragastric pressure drop) after nutrient drink infusion. | Until 2 hours after the start of the liquid meal. Liquid meal started 30 minutes after pancreatic peptide dose or placebo iv infusion.
  Intragastric pressure measurements were assessed using a 36-channel high-resolution solid-state manometry probe. After nutrient drink infusion, the intragastric pressure drops to a minimum value (Nadir), which is a measurement for gastric accommodation, and the pressure restores after. The time point of reaching the Nadir is different between subjects, but pressure is measured until 2 hours after nutrient drink to assess the drop.

SECONDARY OUTCOMES:
The effect of different doses of pancreatic polypeptide infusion on nutrient tolerance. | Infusion of the liquid meal ends after 20 minutes or earlier if max satiation is reached by the subjects.
  Liquid nutrient drink was infused at a constant speed of 60 ml/min. At 1-min intervals subjects were asked to score their satiation using a graphic rating scale that combines verbal descriptors on a scale graded from 0 to 5 (0 is threshold, 5 is maximal satiation. Infusion stopped when the subject reached maximal satiation. The time of infusion is a measurement of their nutrient tolerance.
The effect of different doses of pancreatic polypeptide infusion on gastric emptying rate. | Breath samples were collected in exetainers, twice before and every 15 min after the meal until 6 hours thereafter.
  Gastric emptying rate after placebo and PP 10 pmol/kg*min administration was quantified using the breath test. 13C-labeled sodium octanoate were added to the ND (200 mg/L) and emptying of the stomach was assessed by analysis of the exhaled 13CO2.
The effect of different doses of pancreatic polypeptide infusion on satiety and return of hunger. | Satiety and hunger were scored twice before and every 15 min after the meal until 6 hours thereafter.
  The subjects rate their feeling of satiety (in fasted state)/satiation (in fed state) and hunger using a 100 mm line ranging from 0 to 100, as a response on the questions: 'How hungry do you feel? ' and 'How satisfied do you feel?'. 0 means 'not at all', and 100 means 'extremely much'.
  These feelings cannot be considered to have a better or worse outcome. One expect to have higher hunger and lower satiety scores in fasted state and lower hunger and higher satiation scores in the fed state.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — UZ Leuven
Locations (1):
- Jan Tack, Leuven, Belgium

REFERENCES:
- [Derived] Verbeure W, Rotondo A, Janssen P, Carbone F, Tack J. Supraphysiological effects of pancreatic polypeptide on gastric motor function and nutrient tolerance in humans. Physiol Rep. 2021 Sep;9(17):e15002. doi: 10.14814/phy2.15002. PMID 34435472